CLINICAL TRIAL: NCT06111079
Title: Aspirin Discontinuation at 28 or 36 Weeks' Gestation in High-Risk Pregnant Women of Preeclampsia A Randomized Clinical Trial
Brief Title: Aspirin Discontinuation in High-Risk Pregnant Women of Preeclampsia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: FANG HE (Other)
Responsible Party: Sponsor-Investigator, FANG HE, Chief Physician/Professor of the Obstetrics Department, The Third Affiliated Hospital of Guangzhou Medical University
Organization: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: [2023] Ethics Review NO.118
Record Dates: First submitted 2023-10-23; First posted 2023-11-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Preeclampsia; Perinatal Haemorrhage
Keywords: low dose aspirin; prevention; preeclampsia; pregnancy outcomes; randomized controlled trial; aspirin discontinuation
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: Pregnant women with normal NT scan who meet at least one high-risk factor or at least two medium-risk factors are included. Initiating aspirin 100mg qn during 12-16 weeks of gestation. At 24-27+6 weeks of gestation, the patients were 1:1 randomly divided into two groups. The experimental group discontinue aspirin at 28 weeks of gestation, and the control group receive aspirin until 36 weeks of gestation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin discontinuation group (Experimental): initiation of aspirin 100mg qn from 12 to 16 weeks of gestation, receiving 1:1 randomized grouping at 24-27+6 weeks of gestation, discontinuing aspirin at 28 weeks of gestation.
  Interventions: Drug: aspirin discontinuation
- Control group (Active Comparator): initiation of aspirin 100mg qn from 12 to 16 weeks of gestation, receiving 1:1 randomized grouping at 24-27+6 weeks of gestation, continuing aspirin until 36 weeks of gestation.
  Interventions: Drug: aspirin continuation

INTERVENTIONS:
Drug: aspirin discontinuation — Initiation of aspirin 100mg qn from 12 to 16 weeks of gestation, discontinuing aspirin at 28 weeks of gestation according to randomization at 24-27+6 weeks of gestation.
  Other Names: initiation of aspirin in early pregnancy
  Arms: Aspirin discontinuation group
Drug: aspirin continuation — Initiation of aspirin 100mg qn from 12 to 16 weeks of gestation, continuing aspirin until 36 weeks of gestation according to randomization at 24-27+6 weeks of gestation.
  Other Names: initiation of aspirin in early pregnancy
  Arms: Control group

SUMMARY:
Low-dose aspirin (LDA) is considered to be the most effective agent to prevent preeclampsia (PE). At present, there is little exploration about the timing of aspirin discontinuation. Most international guidelines default until 36 weeks of gestation or delivery. China Guideline (2020) recommended that aspirin should be preventively used until 26-28 weeks of gestation, but there was little direct evidence. According to the two-stage theory, placental dysplasia before 28 weeks of gestation is the key to developing PE, the significance of aspirin use after 28 weeks of gestation is debatable. If aspirin discontinuation at 28 weeks of gestation is proven to be feasible for preventing preterm PE, it will not only reduce the risk of Perinatal Haemorrhage but also save medical expenses.

DETAILED DESCRIPTION:
This study aimed to optimize the strategy of aspirin to prevent preeclampsia, by exploring whether aspirin discontinuation at 28 weeks of gestation to prevent preterm PE is not inferior to 36 weeks of gestation. We will include pregnant women with normal NT scan who meet at least one high-risk factor or at least two medium-risk factors. During 12-16 weeks of gestation, the mean arterial pressure (MAP) and placental growth factor (PlGF) are measured, then initiating aspirin 100mg qn. At 24-27+6 weeks of gestation, the patients were 1:1 randomly divided into two groups, sFlt-1 and PlGF were detected at the same time. The experimental group discontinue aspirin at 28 weeks of gestation, and the control group receive aspirin until 36 weeks of gestation. The incidence of preterm PE in the two groups was compared by non-inferiority test, and the non-inferiority threshold was 2%.

ELIGIBILITY:
Inclusion Criteria:

1. At <16 weeks of gestation, normal NT scan
2. At least 1 high risk factor or at least 2 moderate risk factors
3. Intend to receive prenatal examination and deliver in this institution
4. Signed a written informed consent for participation in the study

Exclusion Criteria:

1. Aspirin initiated after 16 week
2. Intolerant or allergic to aspirin
3. Aspirin adherence was <80%
4. Miscarriage or termination of pregnancy before randomization
5. drop out (do not return to the hospital for delivery).
6. Lost to follow-up

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1800 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of preterm preeclampsia | Within one week after delivery
  delivery with preeclampsia before 37 weeks of gestation

SECONDARY OUTCOMES:
Incidence of early-onset preeclampsia | Within one week after delivery
  delivery with preeclampsia before 34 weeks of gestation
Incidence of term preeclampsia | Within one week after delivery
  delivery with preeclampsia after 37 weeks of gestation
Incidence of gestational hypertension | Within one week after delivery
  new onset of high blood pressure after 20 weeks of gestation (systolic blood pressure ≥140 mm Hg and/or diastolic blood pressure ≥90 mm Hg)
Incidence of small for gestational age | Within one week after delivery
  birth weight below the 10th percentile

CONTACTS AND LOCATIONS:
Overall Officials: Fang He, M.D, Principal Investigator — The Third Affiliated Hospital of Guangzhou Medical University
Locations (1):
- FANG HE, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No